CLINICAL TRIAL: NCT01989871
Title: Adjusted Individual Oral Feeding for Improving Short and Long Term Outcomes of Preterm
Brief Title: Adjusted Individual Oral Feeding for Improving Short and Long Term Outcomes of Preterm Infants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: SHEBA-12-9574-IM-CTIL
Record Dates: First submitted 2013-11-06; First posted 2013-11-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Body Weight Changes; Feeding and Eating Disorders of Childhood; Breast Feeding; Evoked Response Audiometry
Keywords: preterm; oral feeding; outcome
MeSH Terms: conditions — Body Weight Changes; Feeding and Eating Disorders of Childhood; Breast Feeding; Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- protocol feeding (No Intervention): Feeding of preterm infants according to current unit protocol: every 3 hours a prescribed amount
- Adjusted individual feeding (Experimental): Feeding every 2-4 hours, starting with que of hunger and finished upon infant signs.
  Interventions: Behavioral: Adjusted individual feeding

INTERVENTIONS:
Behavioral: Adjusted individual feeding — Feeding every 2-4 hours, starting with ques of hunger and finished upon infant signs.
  Arms: Adjusted individual feeding

SUMMARY:
The authors hypothesize that adjusted individual feeding (AIF) for preterm infant starting from transition to oral feeding (33 weeks corrected age) will result in less episodes of apnea/bradycardia, early achievement of full oral feeding, improved weight gain and shorten hospitalization duration in the short term.

In the long term AIF will result in higher scores on the Griffith's developmental scales, decreasing parental anxiety and feeding disorders .

DETAILED DESCRIPTION:
Preterm infants born at <32 weeks of gestation at our institute will qualify for this study. Recruitment will occur between day 7-14 of life after sever brain malformations or intraventricular bleeding will be ruled out. Randomization to control or intervention will be via sealed envelopes. In the control group - infants will be treated according to the common practice in the neonatal intensive care unit. Transition to oral feeding will occur at 33 wkks (breast feeding) and 34 wks (bottle feeding). Meals will be given every 3 hours, the amount will be written by the care giving physician and will be written as a strict number (i.e 30 ml every 3 hours) Parents in the intervention group will be taught be the nurses (NIDCAP trainees) to identify their infants' ques (self regulation or withdrawn as well as signs of hunger), This parents will be taught the physiology of maturation of feeding, as well as various techniques of infants feeding amongst them pace feeding. During the study parents in both groups will be interviewed every 14 days as for their satisfactions, anxieties, infants ability to cope. video typing during Kangaroo care at 32 and 35 wks as well as during feeding at 35 weeks will be done and evaluated. General movements assessment (neurodevelopment) will be done at 33 -35 weeks gestational age, as well as at 52 weeks. Alberta infant motor scales will be evaluated at 4 and 8 month corrected age,Automated Brain stem evoked Response (ABR) will be done at 33 wks for assessment of brain stem maturity, duration of hospitalization, weight gain per week at 33, 34 and 35 weeks will be calculated, age at full oral feeding will be noted. At the age of 6 month Griffith's developmental scales will be performed

ELIGIBILITY:
Inclusion Criteria:

- birth at less than 32 weeks of gestation

Exclusion Criteria:

* High grade intraventricular hemorrhage (grade 3 or4)
* genetic syndrome

Ages: 25 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
length of hospitalization | between 36-40 weeks gestational age
  length of hospitalization from admission to discharge, and length of stay beyond reaching 36 weeks corrected age , the time point at wich health infants are usually being discharged

SECONDARY OUTCOMES:
age at reaching full oral feedings | between 34-38 gestational age
  the age at which no nasogastric tube was used

OTHER OUTCOMES:
Griffith's developmental scales | 6 month corrected age
  Griffith's developmental scales (Gross and fine motor, speech and language, performance and social skills)
weekly weight gain | 33- 36 weeks gestational age
  weekly weight gain gr/kg will be calculated at 33 weeks gestational age, at 34, 35, and 36 weeks
parental anxiety | 6 month corrected age
  parents anxiety will be assessed by a questioner

CONTACTS AND LOCATIONS:
Overall Officials: Iris Morag, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel